CLINICAL TRIAL: NCT04067141
Title: The Clinical Comparison of the Clariti 1 Day and DAILIES AquaComfort PLUS Daily Disposable Contact Lenses
Brief Title: The Clinical Comparison of Somofilcon A 1 Day and Nelfilcon A Daily Disposable Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: EX-MKTG-75
Record Dates: First submitted 2019-08-21; First posted 2019-08-26 (Actual); Results first posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Ametropia
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Intervention Model Description: This is a bilateral crossover study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- somofilcon A, then nelfilcon A (Experimental): Subjects will bilaterally wear the somofilcon A lenses, then crossover to nelfilcon A lenses after one week of wear. Both lenses will be worn on a daily wear basis for one week.
  Interventions: Device: somofilcon A; Device: nelfilcon A
- nelfilcon A, then somofilcon A (Experimental): Subjects will bilaterally wear the nelfilcon A lenses, then crossover to somofilcon A lenses after one week of wear. Both lenses will be worn on a daily wear basis for one week.
  Interventions: Device: somofilcon A; Device: nelfilcon A

INTERVENTIONS:
Device: somofilcon A — Contact Lens
  Other Names: somofilcon A 1 day; test lens; clariti 1 day
Device: nelfilcon A — Contact Lens
  Other Names: nelfilcon A Daily Disposable Contact Lens; control lens; DAILIES AquaComfort PLUS daily disposable

SUMMARY:
This subject-masked, randomized, bilateral crossover study will compare the clinical performance and subjective acceptance of the somofilcon A 1 day soft contact lens with the nelfilcon A daily disposable lens when used on a daily wear, daily disposable basis.

DETAILED DESCRIPTION:
This will be a randomized, subject-masked, crossover, bilateral study, controlled by cross-comparison. This will compare the clinical performance and subjective acceptance of the somofilcon A 1 day soft contact lens with the nelfilcon A daily disposable lens when used on a daily wear, daily disposable basis.

Subjects will use each lens type for a week in random sequence. Follow-up visits for each lens will be performed after one week of wear. Lenses will be worn on a daily wear, daily disposable wear schedule.

ELIGIBILITY:
Inclusion Criteria:

* They are of legal age (18) and capacity to volunteer.
* They understand their rights as a research subject and are willing and able to sign a Statement of Informed Consent.
* They are willing and able to follow the protocol.
* They agree not to participate in other clinical research for the duration of this study.
* They have a contact lens spherical prescription between -1.00 to - 6.00D (inclusive)
* They have a maximum of -1.00DC ocular astigmatism in each eye.
* They can be satisfactorily fitted with the study lens types.
* At dispensing, they can attain at least 0.20 logMAR distance high contrast visual acuity in each eye with the study lenses within the available power range.
* They currently use soft contact lenses or have done so in the previous six months.
* They are willing to comply with the wear schedule (at least five days per week and for at least eight hours per day).
* They own a wearable pair of spectacles.

Exclusion Criteria:

* They have an ocular disorder which would normally contra-indicate contact lens wear.
* They have a systemic disorder which would normally contra-indicate contact lens wear.
* They are using any topical medication such as eye drops or ointment.
* They have had cataract surgery.
* They have had corneal refractive surgery.
* They have any corneal distortion resulting from previous hard or rigid lens wear or have keratoconus.
* They are pregnant or breast-feeding.
* They have any ocular abnormality which would, in the opinion of the investigator, normally contraindicate contact lens wear.
* They have any infectious disease which would, in the opinion of the investigator, contraindicate contact lens wear or pose a risk to study personnel, or they have any immunosuppressive disease (e.g. HIV), or a history of anaphylaxis or severe allergic reaction.
* They have taken part in any other contact lens or care solution clinical trial or research, within two weeks prior to starting this study.
* They currently wear either the clariti 1day or the DAILIES AquaComfort Plus lens.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-07-04 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2019-11-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Eurolens Research, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: First Intervention
Arm/Group | Somofilcon A, Then Nelfilcon A | Nelfilcon A, Then Somofilcon A
Started | 35 | 35
Completed | 35 | 34
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Second Intervention
Arm/Group | Somofilcon A, Then Nelfilcon A | Nelfilcon A, Then Somofilcon A
Started | 34 (Unacceptable lens fit at dispense. One withdrawal by subject.) | 33 (Unacceptable lens fit at dispense. One withdrawal by subject)
Completed | 34 | 31
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Subjects were randomized to wear somofilcon A 1 day and nelfilcon A for one week in this cross-over study.
Arm/Group | Overall Study
Number analyzed (Participants) | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 70
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.6 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 70

OUTCOME MEASURES:

1. Primary Outcome: Subjective Comfort at Lens Dispensing
Description: Subjective comfort at lens dispensing on scale 0-100 (0=Causes pain. Cannot be tolerated to 100=Excellent. Cannot be felt.).
Time Frame: Baseline (after 5 minutes of lens dispense)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Somofilcon A: Subjects will bilaterally wear the somofilcon A lenses for 1 week.
  somofilcon A: Contact Lens
- Nelfilcon A: Subjects will bilaterally wear the nelfilcon A lenses for 1 week.
  nelfilcon A: Contact Lens
Arm/Group | Somofilcon A | Nelfilcon A
Number analyzed (Participants) | 69 | 69
units on a scale | 90.9 (11.6) | 88.5 (12.8)

2. Primary Outcome: Subjective Comfort at Start of Day
Description: Subjective comfort at start of day on scale 0-100 (0=Causes pain. Cannot be tolerated to 100=Excellent. Cannot be felt.).
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A | Nelfilcon A
Number analyzed (Participants) | 67 | 68
units on a scale | 89.9 (13.8) | 87.0 (14.7)

3. Primary Outcome: Subjective Comfort at End of Day
Description: Subjective comfort at end of day on scale 0-100 (0=Causes pain. Cannot be tolerated to 100=Excellent. Cannot be felt.).
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A | Nelfilcon A
Number analyzed (Participants) | 67 | 68
units on a scale | 75.9 (22.1) | 68.0 (25.5)

4. Primary Outcome: Overall Subjective Comfort
Description: Overall subjective comfort on scale 0-100 (0=Causes pain. Cannot be tolerated to 100=Excellent. Cannot be felt.).
Time Frame: Baseline (after 5 minutes of lens dispense)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A | Nelfilcon A
Number analyzed (Participants) | 69 | 69
units on a scale | 90.4 (10.1) | 90.9 (10.8)

5. Primary Outcome: Overall Subjective Comfort
Description: Overall subjective comfort on scale 0-100 (0=Causes pain. Cannot be tolerated to 100=Excellent. Cannot be felt.).
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A | Nelfilcon A
Number analyzed (Participants) | 67 | 68
units on a scale | 86.1 (14.1) | 78.8 (19.8)

6. Primary Outcome: Subjective Vision
Description: Subjective Vision rated on scale 0-100 (0=unacceptable, lens cannot be worn to 100=excellent, unaware of an visual loss.)
Time Frame: Baseline (after 5 minutes of lens dispense)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A | Nelfilcon A
Number analyzed (Participants) | 69 | 69
units on a scale | 92.8 (10.1) | 94.2 (7.8)

7. Primary Outcome: Subjective Vision
Description: as for outcome 6
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A | Nelfilcon A
Number analyzed (Participants) | 67 | 68
units on a scale | 90.9 (12.1) | 92.1 (13.2)

8. Secondary Outcome: Biomicroscopy - Conjunctival Redness Score
Description: Conjunctival redness - slit lamp biomicroscopy using Efron Grading Scale, 0 - 4 (0=normal, 1=trace, 2=mild, 3=moderate, 4=severe).
Time Frame: One Week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A | Nelfilcon A
Number analyzed (Participants) | 67 | 68
units on a scale | 0.85 (0.25) | 0.87 (0.25)

9. Secondary Outcome: Biomicroscopy - Limbal Redness Score
Description: Limbal redness - slit lamp biomicroscopy using Efron Grading Scale, 0 - 4 (0=normal, 1=trace, 2=mild, 3=moderate, 4=severe).
Time Frame: One week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A | Nelfilcon A
Number analyzed (Participants) | 67 | 68
units on a scale | 0.74 (0.27) | 0.79 (0.28)

10. Secondary Outcome: Biomicroscopy - Corneal Staining Score
Description: Corneal staining - slit lamp biomicroscopy using Efron Grading Scale, 0 - 4 (0=normal, 1=trace, 2=mild, 3=moderate, 4=severe).
Time Frame: One week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A | Nelfilcon A
Number analyzed (Participants) | 67 | 68
units on a scale | 0.33 (0.43) | 0.32 (0.40)

11. Secondary Outcome: Biomicroscopy - Conjunctival Staining Score
Description: Conjunctival staining - slit lamp biomicroscopy using Efron Grading Scale, 0 - 4 (0=normal, 1=trace, 2=mild, 3=moderate, 4=severe).
Time Frame: One week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A | Nelfilcon A
Number analyzed (Participants) | 67 | 68
units on a scale | 1.46 (0.71) | 0.35 (0.36)

12. Secondary Outcome: Biomicroscopy - Papillary Conjunctivitis Score
Description: Papillary conjunctivitis- slit lamp biomicroscopy using Efron Grading Scale, 0 - 4 (0=normal, 1=trace, 2=mild, 3=moderate, 4=severe).
Time Frame: One week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A | Nelfilcon A
Number analyzed (Participants) | 67 | 68
units on a scale | 1.02 (0.20) | 1.03 (0.18)

13. Secondary Outcome: Horizontal Centration - Lens Fit
Description: Horizontal centration graded by -2 to 2 (-2= Extremely nasal, -1 slightly nasal, 0=optimum, 1=slightly temporal, 2=extremely temporal).
Time Frame: Baseline (after 5 minutes of lens dispense)
Measure: Number; unit: percentage of lenses
Arm/Group | Somofilcon A | Nelfilcon A
Number analyzed (Participants) | 69 | 70
percentage of lenses
  Extremely nasal | 0 | 0
  Slightly nasal | 6 | 6
  Optimum | 51 | 63
  Slightly temporal | 43 | 31
  Extremely temporal | 0 | 0

14. Secondary Outcome: Horizontal Centration - Lens Fit
Description: as for outcome 13
Time Frame: One Week
Measure: Number; unit: percentage of lenses
Units Other Than Participants: eyes
Arm/Group | Somofilcon A | Nelfilcon A
Number analyzed (Participants) | 66 | 68
Number analyzed (eyes) | 132 | 136
percentage of lenses
  Extremely nasal | 0 | 0
  Slightly nasal | 3 | 1
  Optimum | 41 | 57
  Slightly temporal | 56 | 41
  Extremely temporal | 0 | 0

15. Secondary Outcome: Vertical Centration Grade - Lens Fit
Description: Vertical centration graded by -2 to 2 (-2= Extremely inferior, -1 slightly inferior, 0=optimum, 1=slightly superior, 2=extremely superior).
Time Frame: Baseline (after 5 minutes of lens dispense)
Measure: Number; unit: percentage of lenses
Units Other Than Participants: eyes
Arm/Group | Somofilcon A | Nelfilcon A
Number analyzed (Participants) | 69 | 70
Number analyzed (eyes) | 138 | 140
percentage of lenses
  Extremely inferior | 1 | 0
  Slightly inferior | 17 | 43
  Optimum | 49 | 49
  Slightly superior | 32 | 9
  Extremely superior | 0 | 0

16. Secondary Outcome: Vertical Centration Grade - Lens Fit
Description: as for outcome 15
Time Frame: One week
Measure: Number; unit: percentage of lenses
Units Other Than Participants: eyes
Arm/Group | Somofilcon A | Nelfilcon A
Number analyzed (Participants) | 66 | 68
Number analyzed (eyes) | 132 | 136
percentage of lenses
  Extremely inferior | 0 | 0
  Slightly inferior | 23 | 50
  Optimum | 44 | 44
  Slightly superior | 33 | 6
  Extremely superior | 0 | 0

17. Secondary Outcome: Corneal Coverage Grade
Description: Corneal coverage graded by -2 to 2 (-2=extremely inadequate, -1=slightly inadequate, but acceptable, 0=optimum, 1=slightly excessive, but acceptable, 2=extremely excessive).
Time Frame: Baseline (after 5 minutes of lens dispense)
Measure: Number; unit: percentage of lenses
Units Other Than Participants: eyes
Arm/Group | Somofilcon A | Nelfilcon A
Number analyzed (Participants) | 69 | 70
Number analyzed (eyes) | 138 | 140
percentage of lenses
  Extremely inadequate | 1 | 0
  Slightly inadequate | 28 | 23
  Optimum | 71 | 74
  Slightly excessive | 0 | 3
  Extremely excessive | 0 | 0

18. Secondary Outcome: Corneal Coverage Grade
Description: as for outcome 17
Time Frame: One week
Measure: Number; unit: percentage of lenses
Units Other Than Participants: eyes
Arm/Group | Somofilcon A | Nelfilcon A
Number analyzed (Participants) | 66 | 68
Number analyzed (eyes) | 132 | 136
percentage of lenses
  Extremely inadequate | 0 | 1
  Slightly inadequate | 36 | 26
  Optimum | 64 | 71
  Slightly excessive | 0 | 1
  Extremely excessive | 0 | 0

19. Secondary Outcome: Post-Blink Movement Grade
Description: Post-blink movement graded by -2 to 2 (-2=extremely inadequate, -1=slightly inadequate, but acceptable, 0=optimum, 1=slightly excessive, but acceptable, 2=extremely excessive).
Time Frame: Baseline (after 5 minutes of lens dispense)
Measure: Number; unit: percentage of lenses
Units Other Than Participants: eyes
Arm/Group | Somofilcon A | Nelfilcon A
Number analyzed (Participants) | 69 | 70
Number analyzed (eyes) | 138 | 140
percentage of lenses
  Extremely inadequate | 0 | 0
  Slightly inadequate | 17 | 19
  Optimum | 65 | 57
  Slightly Excessive | 16 | 24
  Extremely Excessive | 1 | 0

20. Secondary Outcome: Post-Blink Movement Grade
Description: as for outcome 19
Time Frame: 1 week
Measure: Number; unit: percentage of lenses
Units Other Than Participants: eyes
Arm/Group | Somofilcon A | Nelfilcon A
Number analyzed (Participants) | 66 | 68
Number analyzed (eyes) | 132 | 136
percentage of lenses
  Extremely inadequate | 0 | 0
  Slightly inadequate | 21 | 26
  Optimum | 67 | 46
  Slightly Excessive | 12 | 26
  Extremely Excessive | 0 | 1

21. Secondary Outcome: Ocular Redness Rating
Description: Ocular redness rating rated on a scale 0-100 (0=extremely poor, intolerable levels of redness to 100 = excellent, no redness)
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A | Nelfilcon A
Number analyzed (Participants) | 67 | 68
units on a scale | 94.1 (8.9) | 92.8 (12.7)

ADVERSE EVENTS:
Time Frame: From dispense up to 1 week on each study lens for a total of two weeks.
Arm/Group | Somofilcon A | Nelfilcon A
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/70
Other Adverse Events (participants affected / at risk) | 2/70 | 0/70
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Somofilcon A (N=70) | Nelfilcon A (N=70)
Bacterial conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Corneal Abrasion (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-06): https://cdn.clinicaltrials.gov/large-docs/41/NCT04067141/Prot_SAP_000.pdf